CLINICAL TRIAL: NCT06426745
Title: Split-dose Versus Single-dose Bowel Preparation for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PEG solution
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Colonic Cancer; Colonic Polyp; IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps; Irritable Bowel Syndrome | interventions — Cathartics; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split-dose bowel preparation (Experimental): About 90 participants underwent Split-dose bowel preparation for colonoscopy
  Interventions: Procedure: Bowel preparation
- single-dose bowel preparation (Experimental): About 90 participants underwent single-dose bowel preparation for colonoscopy
  Interventions: Procedure: Bowel preparation

INTERVENTIONS:
Procedure: Bowel preparation — to compare bowel cleanliness, compliance, tolerability, and patient satisfaction of a single regimen versus a split regimen for colonoscopy.
  Other Names: colonoscopy

SUMMARY:
Colonoscopy is the current standard method for evaluation of colonic disorders such as colorectal cancer, IBD, polyps, and other conditions.

DETAILED DESCRIPTION:
Colonic cancers are a major concern in the Middle East and the world in general, and every institute has attempted to initiate various clinical and investigatory procedures to detect the disease early in its development. From 2005 till 2010 an audit conducted at the Royal Liverpool University revealed that out of 8910 colonoscopies, 693 were incomplete (7.8%), and for 25% of failure was because of inadequate bowel preparation.

An adequate bowel preparation regimen is not only effective in cleansing the colon but should be well tolerated by patients. The polyethylene glycol (PEG) solution, an isosmotic non-absorbable polymer, is generally used for bowel preparation, because of its safety, effectiveness, and good tolerability. Quality of bowel cleansing depends not only on the formula used, but the preparation regimen also plays a role. Split dosing of the laxative offers, in general, better cleansing than a single dose preparation.

A large survey was also done in the USA in 2018 and demonstrated that split dose treatment was more tolerable than single-dose treatment for bowel preparation.

Also more recent study shows split-dose bowel preparation for colonoscopy with PEG is better than single-dose, in terms of adequate bowel preparation and polyp detection.

On the other hand , a large randomized trial of PEG regimens show, low-volume same-day resulted in similar bowel cleanliness compared with high-volume or low-volume split-dosing. Willingness to repeat and tolerability were superior with low-volume same-day compared with high-volume split-dose and similar to low-volume split-dose. Another most recent one demonstrated that same-day morning PEG regimen can be considered an effective well-tolerated, and acceptable bowel preparation for colonoscopy.

A same-day dose of bowel cleanser has several benefits compared with split-dose or previous-day dose: the fasting time is shorter and there is no sleep disturbance, which can be associated with split-dose or previous-day regimen.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing elective colonoscopy

Exclusion Criteria:

* Presence of sever renal impairment. (Creatinine clearance < 30 ml/min or patient on hemodialysis).
* Sever congestive heart failure (NHYA III or IV).
* Pregnant woman.
* History of bowel obstruction or resection.
* Known allergies to polyethylene glycol.
* Refusal of consent for the study.
* Signs of liver cell failure as ascites and hepatic encephalopathy.
* Electrolytes disturbances

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
colon cleansing | 2 hours before Bowel Preparation
  to compare the efficacy of split-dose versus single morning administration of PEG solution for colon cleansing in patient undergoing colonoscopy using Boston Bowel Preparation Scale , and to assess the optimal preparation- to-colonoscopy (PC) interval .

CONTACTS AND LOCATIONS:
Overall Officials: Seham Mohammad Abd-AlAdl Seif, Professor, Study Chair — Internal Medicine Hepatology and Gastroenterology Faculty of Medicine - Mansoura University; Hany Shabana, M.D, Study Director — Hepatology and Gastroenterology Faculty of Medicine - Mansoura University
Locations (1):
- Mansoura university Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No